CLINICAL TRIAL: NCT03037775
Title: The Influence of Electronic and Traditional Cigarettes Smoking on Hemodynamic Parameters and Sympathetic Nerves Activity in Healthy People
Brief Title: The Influence of Electronic and Traditional Cigarettes Smoking on Hemodynamic Parameters
Acronym: EPAPHemo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Jacek Lewandowski, M.D., Ph.D., Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EPAPHemo
Record Dates: First submitted 2017-01-11; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Tobacco; Use, Harmful
Keywords: tobacco; cardiovascular system; sympathetic nervous system
MeSH Terms: interventions — BaseLine dental cement; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigated group (Other): Subjects underwent procedures: hemodynamic indices will be measured at baseline and during 1/ e-cigarette without nicotine smoking, 2/ e-cigarette with nicotine and during 3/ traditional cigarette smoking in random order
  Interventions: Other: Baseline; Device: e-cigarette without nicotine; Device: e-cigarette with nicotine; Device: traditional cigarette

INTERVENTIONS:
Other: Baseline — measurement of baseline hemodynamic parameters
Device: e-cigarette without nicotine — measurement hemodynamic parameters during smoking e-cigarette without nicotine
Device: e-cigarette with nicotine — measurement hemodynamic parameters smoking e-cigarette with nicotine
Device: traditional cigarette — measurement hemodynamic parameters smoking traditional cigarette

SUMMARY:
It is intended to examine 50 healthy volunteers aged 18 - 60 years. 12-hour abstinence from tobacco smoke, alcohol or coffee before the experiment will be required. The exclusion criteria are medical history of stroke, coronary artery disease, chronic heart failure, hypertension, peripheral vascular disease, atrial fibrillation, polyneuropathy, obesity (BMI> 30 kg/m2), the current active disease (eg. viral infection). Test subjects will actively inhale for 10 minutes tobacco or the e-cigarette smoke with nicotine fluid (18 mg/ml) or fluid without nicotine for 10 minutes. The study protocol involves random allocation to groups exposed to electronic or traditional cigarette smoke in cross-over scheme. The primary endpoint is the maximum change in heart rate compared to mean values prior to exposure. Secondary end points is the maximum change in the measured parameters (hemodynamic and autonomic values) compared to the average values before exposure. The measurements will be performed using the Task Force Monitor system for non-invasive measurement of hemodynamic parameters and the assessment of autonomic function. Adrenergic activity will be tested with microneurography. A periodic analysis is planned after examining 15 and 35 patients.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers aged 18 - 60 years
* 12-hour abstinence from tobacco smoke, alcohol or coffee before the experiment will be required

Exclusion Criteria:

* history of stroke, coronary artery disease, chronic heart failure, hypertension, peripheral vascular disease, atrial fibrillation, polyneuropathy, obesity (BMI> 30 kg/m2), the current active disease (eg. viral infection).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | through study completion, an average of 1 year
  RR intervals in ms, very low frequency (VLF), low frequency (LF), and high frequency (HF) components - ms2

SECONDARY OUTCOMES:
Systolic, diastolic, mean blood pressure | through study completion, an average of 1 year
  mm Hg
Heart rate | through study completion, an average of 1 year
  beats/min
Blood pressure variability | through study completion, an average of 1 year
  mm Hg
Puls wave velocity | through study completion, an average of 1 year
  m/s
Stroke Volume | through study completion, an average of 1 year
  ml
Cardiac output | through study completion, an average of 1 year
  ml/min
Total Peripheral Resistance | through study completion, an average of 1 year
  dyn*sec/cm5
Baroreceptor reflex sensitivity | through study completion, an average of 1 year
  ms/mm Hg
Muscle sympathetic nerve activity | through study completion, an average of 1 year
  bursts/min, bursts/100 beats/min

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Lewandowski, M.D., Ph.D., Principal Investigator — Medical University of Warsaw
Locations (1):
- Warszawski Uniwersytet Medyczny, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No